CLINICAL TRIAL: NCT04598451
Title: A Randomized, Double-Blinded, Placebo-Controlled Trial to Investigate the Efficacy, Safety, and Tolerability of Efgartigimod PH20 SC in Adult Patients With Pemphigus (Vulgaris or Foliaceus)
Brief Title: A Study to Assess the Efficacy and Safety of a Subcutaneous Formulation of Efgartigimod PH20 SC in Adults With Pemphigus (Vulgaris or Foliaceus)
Acronym: ADDRESS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARGX-113-1904
Record Dates: First submitted 2020-10-08; First posted 2020-10-22 (Actual); Results first posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Pemphigus Vulgaris; Pemphigus Foliaceus
MeSH Terms: conditions — Pemphigus | interventions — Prednisone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- efgartigimod PH20 SC (Experimental): patients receiving efgartigimod PH20 SC on top of prednisone
  Interventions: Biological: efgartigimod PH20 SC; Drug: prednisone
- placebo (Experimental): patients receiving placebo on top of prednisone
  Interventions: Other: Placebo; Drug: prednisone

INTERVENTIONS:
Biological: efgartigimod PH20 SC — Subcutaneous injection of efgartigimod using rHuPH20 (PH20) as a permeation enhancer
  Arms: efgartigimod PH20 SC
Other: Placebo — Subcutaneous injection of placebo
  Arms: placebo
Drug: prednisone — Oral prednisone tablets

SUMMARY:
This is a prospective, multicenter, randomized, double-blinded, placebo-controlled trial to investigate the efficacy, safety, patient outcome measures, tolerability, immunogenicity, PK, and PD of efgartigimod PH20 SC in adult participants aged from 18 years with PV or PF. The trial comprises a screening period of up to 3 weeks, a treatment period of up to 30 weeks, and an 8-week follow-up period for participants who do not enroll into the open-label extension (OLE) trial ARGX-113-1905. The primary objective of the ARGX-113-1904 trial is to demonstrate the efficacy of subcutaneous administration of efgartigimod co-formulated with recombinant human hyaluronidase PH20 (Efgartigimod PH20 SC) compared to placebo in the treatment of participants with Pemphigus Vulgaris (PV). Secondary objectives are to also demonstrate the efficacy of efgartigimod PH20 SC in the treatment of participants with Pemphigus Foliaceus (PF), and to demonstrate early onset of action and a prednisone-sparing effect. After confirmation of eligibility, participants will be randomized in a 2: 1 ratio to receive efgartigimod PH20 SC or placebo

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the requirements of the trial, to provide written informed consent (including consent for the use and disclosure of research-related health information), willingness and ability to comply with the trial protocol procedures (including required trial visits).
2. The participant is male or female, and aged from 18 years at the time of signing the informed consent form (ICF).
3. The participant has a clinical diagnosis of PV (mucosal, cutaneous, mucocutaneous) or PF which has been confirmed by cutaneous histology, positive direct immunofluorescence (IF), and positive indirect IF and/or enzyme-linked immunosorbent assay (ELISA).
4. The participant meets one of the following profiles:

   1. Newly diagnosed disease with PDAI ≥15 at baseline and naïve to treatment
   2. Newly diagnosed disease with PDAI ≥15 while receiving a first course of oral prednisone (or equivalent). According to clinical judgment, the participant has shown no significant improvement of PV or PF signs for at least 2 weeks before baseline and is considered fit to start prednisone treatment at 0.5 mg/kg qd at baseline.
   3. Experiencing flare with PDAI ≥15, a maximum of 4 years since diagnosis, and off prednisone therapy ± a conventional immunosuppressant (e.g., azathioprine, cyclophosphamide, methotrexate, mycophenolate mofetil) or dapsone. Note: conventional immunosuppressants and dapsone must be discontinued before baseline.
   4. Experiencing flare with PDAI ≥15, a maximum of 4 years since diagnosis, and receiving a tapered dose of oral prednisone (or the equivalent), provided that prednisone has been given at stable dose ± a conventional immunosuppressant for at least 2 weeks and patients are fit to start prednisone treatment at 0.5 mg/kg qd at baseline.
5. Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating clinical trials and:

   1. Male participants: Male participants must agree to use acceptable method of contraception, and not donate sperm from signing the ICF until the end of the study.
   2. Female participants: Women of childbearing potential must:

      * have a negative serum pregnancy test at screening and negative urine pregnancy test at baseline before the IMP can be administered.
      * agree to use a highly effective or acceptable contraception method, which should be maintained at minimum until after the last dose of IMP
6. For Japanese participants enrolled in sites in Japan only: A Japanese participant is defined as a participant whose parents and 4 grandparents are Japanese, and who has Japanese nationality, was born in Japan, has not lived outside of Japan for a total of >10 years, and currently lives in Japan.

Exclusion Criteria:

1. Participant has a confirmed diagnosis of paraneoplastic pemphigus, drug-induced pemphigus, pemphigus vegetans, pemphigus erythematosus, or any other non-PV/non-PF autoimmune blistering disease.
2. Participants with mild disease severity as defined by PDAI <15 at baseline.
3. Participants who show a significant improvement of PV or PF in the period from screening to baseline according to clinical judgment (eg, the patient has achieved DC or a substantial reduction in PDAI activity score during screening period).
4. The participant has been administered therapy(ies) other than oral prednisone or conventional immunosuppressants (e.g., azathioprine, cyclophosphamide, methotrexate, mycophenolate mofetil) or dapsone within 2 months before the baseline visit and that can affect clinical disease activity. For example, excluded medications are intravenous methylprednisolone, dapsone, sulfasalazine, tetracyclines, nicotinamide at doses above the recommended daily allowance (RDA)/dietary reference intake (DRI), plasmapheresis/ plasma exchange, immunoadsorption, and IVIg.
5. Use of any monoclonal antibody (including rituximab or another anti-CD20 biologic) within 6 months before the baseline visit.
6. Known hypersensitivity to any of the components of the administered treatments.
7. The participant has a known contraindication to oral prednisone.
8. The participant has a history of refractory disease, as defined by a failure to respond to first-line and second-line therapies
9. Participants who have a history of malignancy unless deemed cured by adequate treatment with no evidence of recurrence for ≥3 years before first IMP administration. Participants with any of the following cancers can be included at any time, provided they are adequately treated prior to their participation in the study:

   * Basal cell or squamous cell skin cancer,
   * Carcinoma in situ of the cervix,
   * Carcinoma in situ of the breast,
   * Incidental histological finding of prostate cancer
10. Participants with clinical evidence of other significant serious disease or participants who recently underwent or have planned a major surgery during the period of the trial, or any other condition in the opinion of the investigator, that could confound the results of the trial or put the patient at undue risk.
11. Pregnant and lactating women and those intending to become pregnant during the trial.
12. Current or history (i.e. within 12 months of screening) of alcohol, drug, or medication abuse.
13. Any other known autoimmune disease that, in the opinion of the investigator, would interfere with an accurate assessment of clinical symptoms of PV or PF or put the participant at undue risk.
14. The participant has a Karnofsky Performance score <60%.
15. Vaccination with live viral vaccines within 28 days prior to randomization.
16. The participant has clinically significant uncontrolled active or chronic bacterial, viral, or fungal infection.
17. Positive serum test at screening for an active viral infection with any of the following conditions: Hepatitis B Virus, Hepatitis C Virus , HIV.
18. The participant has total immunoglobulin G (IgG) <6 g/L at screening.
19. The participant has previously participated in a trial with efgartigimod and has received at least one administration of IMP.
20. Use of an investigational drug within 3 months or 5 half-lives of the drug (whichever is longer) prior to first IMP administration

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-08-22 (Actual); Study Completion 2023-08-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (134):
- United States (21):
  - Investigator site 77 - US0010086, Birmingham, Alabama
  - Investigator site 97 - US0010091, Scottsdale, Arizona
  - Investigator site 121 - US0010092, Redwood City, California
  - Investigator site 125 - US0010153, Castle Rock, Colorado
  - Investigator site 2 - US0010087, Boca Raton, Florida
  - Investigator site 99 - US0010117, Miami, Florida
  - Investigator site 78 - US0010109, Orlando, Florida
  - Investigator site 127 - US0010155, West Lafayette, Indiana
  - Investigator site 61 - US0010090, Minneapolis, Minnesota
  - Investigator site 102 - US0010098, St Louis, Missouri
  - Investigator site 19 - US0010088, Buffalo, New York
  - Investigator site 136 - US0010196, New York, New York
  - Investigator site 60 - US0010096, Durham, North Carolina
  - Investigator site 20 - US0010094, Cleveland, Ohio
  - Investigator site 73 - US00100, Philadelphia, Pennsylvania
  - Investigator site 101 - US0010097, Philadelphia, Pennsylvania
  - Investigator site 98 - US0010107, Dallas, Texas
  - Investigator site 1 - US0010084, Dripping Springs, Texas
  - Investigator site 126 - US0010182, Houston, Texas
  - Investigator site 88 - US0010114, Houston, Texas
  - Investigator site 59 - US0010106, Norfolk, Virginia
- Australia (3):
  - Investigator site 24 - AU0610006, Sydney, New South Wales
  - Investigator site 5 - AU0610007, Parkville, Victoria
  - Investigator site 103 - AU0610013, Melbourne
- Bulgaria (5):
  - Investigator site 30 - BG350012, Pleven
  - Investigator site 31 - BG3590013, Plovdiv
  - Investigator site 4 - BG3590010, Sofia
  - Investigator site 2 - BG3590009, Sofia
  - Investigator site 13 - BG3590011, Sofia
- China (13):
  - Investigator site 110 - CN0860017, Beijing
  - Investigator site 111 - CN0860018, Chendu
  - Investigator site 131 - CH0860027, Chongqing
  - Investigator site 118 - CN0860023, Fujian
  - Investigator site 120 - CN0860022, Guangzhou
  - Investigator site 128 - CH0860053, Guangzhou
  - Investigator site 109 - CN0860021, Guanzhou
  - Investigator site 119 - CN0860024, Nanjing
  - Investigator site 112 - CN0860020, Shanghai
  - Investigator site 108 - CN0860016, Shanghai
  - Investigator site 113 - CN0860025, Wuhan
  - Investigator site 123 - CN0860019, Wuhan
  - Investigator site 129 - CH0860026, Zhengzhou
- France (4):
  - Investigator site 34 - FR0330028, Bobigny
  - Investigator site 33 - FR0330027, La Tronche
  - Investigator site 46 - FR0330029, Rouen
  - Investigator site 32 - FR0330026, Saint-Etienne
- Georgia (4):
  - Investigator site 63 - GE9950014, Tbilisi
  - Investigator site 132 - GE9950030, Tbilisi
  - Investigator site 35 - GE9950013, Tbilisi
  - Investigator site 36 - GE9950015, Tbilisi
- Germany (10):
  - Investigator site 64 - DE0490029, Berlin
  - Investigator site 48 - DE0490030, Dresden
  - Investigator site 49 - DE0490024, Frankfurt am Main
  - Investigator site 47 - DE0490023, Freiburg im Breisgau
  - Investigator site 38 - DE0490028, Kiel
  - Investigator site 37 - DE0490002, Lübeck
  - Investigator site 68 - DE0490001, Marburg
  - Investigator site 25 - DE0490025, Tübingen
  - Investigator site 79 - DE0490027, Ulm
  - Investigator site 21 - DE0490026, Würzburg
- Greece (6):
  - Investigator site 40 - GR0300004, Athens
  - Investigator site 51 - GR0300006, Athens
  - Investigator site 69 - GR0300001, Athens
  - Investigator site 39 - GR0300003, Chaïdári
  - Investigator site 50 - GR0300002, Thessaloniki
  - Investigator site 41 - GR0300005, Thessaloniki
- Hungary (4):
  - Investigator site 133 - HU0360023, Budapest
  - Investigator site 22 - HU0360003, Debrecen
  - Investigator site 14 - HU0360001, Pécs
  - Investigator site 42 - HU0360002, Szeged
- India (4):
  - Investigator site 80 - IN0910002, Ahmedabad
  - Investigator site 100 - IN0910001, Chandigarh
  - Investigator site 90 - IN0910004, Lucknow
  - Investigator site 91 - IN0910003, Nagpur
- Investigator site 12 - ISR9720002, Tel Aviv, Israel
- Italy (7):
  - Investigator site 11 - IT0390006, Rome, Lazio
  - Investigator site 104 - IT0390039, Catania
  - Investigator site 52 - IT0390031, Florence
  - Investigator site 92 - IT0390030, Genova
  - Investigator site 70 - IT0390038, Perugia
  - Investigator site 43 - IT390005, Roma
  - Investigator site 71 - IT0390040, Siena
- Japan (10):
  - Investigator site 94 - JP0810046, Aichi
  - Investigator site 81 - JP0810040, Hiroshima
  - Investigator site 82 - JP0810042, Kofu
  - Investigator site 85 - JP0810050, Kurume
  - Investigator site 84 - JP0810047, Okayama
  - Investigator site 93 - JP0810041, Okayama
  - Investigator site 86 - JP0810049, Osaka
  - Investigator site 74 - JP0810045, Sapporo
  - Investigator site 124 - JP0810067, Sendai
  - Investigator site 83 - JP0810043, Tokyo
- Poland (5):
  - Investigator site 26 - PL0480027, Katowice
  - Investigator site 72 - PL0480032, Lodz
  - Investigator site 95 - PL0480036, Poznan
  - Investigator site 27 - PL0480025, Rzeszów
  - Investigator site 28 - PL0480028, Wroclaw
- Romania (3):
  - Investigator site 106 - RO0400013, Bucharest
  - Investigator site 105 - RO0400014, Cluj-Napoca
  - Investigator site 107 - RO0400015, Iași
- Russia (8):
  - Investigator site 54 - RU0070035, Chelyabinsk
  - Investigator site 57 - RU0070029, Kazan'
  - Investigator site 55 - RU0070030, Krasnodar
  - Investigator site 53 - RU0070032, Rostov-on-Don
  - Investigator site 56 - RU0070031, Saint Petersburg
  - Investigator site 65 - RU0070034, Saint Petersburg
  - Investigator site 66 - RU0070028, Saratov
  - Investigator site 58 - RU0070033, Yekaterinburg
- Serbia (4):
  - Investigator site 116 - RS3810011, Belgrade
  - Investigator site 122 - RS3810010, Belgrade
  - Investigator site 115 - RS3810012, Niš
  - Investigator site 114 - RS3810009, Novi Sad
- Spain (10):
  - Investigator site 29 - ES0340026, Barcelona
  - Investigator site 15 - ES0340032, Barcelona
  - Investigator site 130 - ES0340053, Granada
  - Investigator site 67 - ES0340034, Madrid
  - Investigator site 10 - ES0340025, Madrid
  - Invetistigator site 8 - ES0340029, Madrid
  - Investigator site 6 - ES0340027, Madrid
  - Investigator site 134 - ES0340057, Málaga
  - Investigator site 23 - ES0340031, Pamplona
  - Investigator site 7 - ES0340028, Seville
- Turkey (Türkiye) (3):
  - Investigator site 76 - TR0900020, Gaziantep
  - Investigator site 75 - TR0900012, Istanbul
  - Investigator site 87 - TR0900011, Istanbul
- Ukraine (6):
  - Investigator site 89 - UA3800017, Dnipro
  - Investigator site 45 - UA3800023, Ivano-Frankivsk
  - Investigator site 16 - UA3800020, Kyiv
  - Investigator site 18 - UA3800019, Kyiv
  - Investigator site 62 - UA3800021, Lviv
  - Investigator site 17 - UA3800018, Zaporizhzhia
- United Kingdom (3):
  - Investigator site 117 - UK0440021, Birmingham
  - Investigator site 96 - UK0440022, Bristol
  - Investigator site 135 - GB0440037, Southampton

RESULTS

PARTICIPANT FLOW:
Groups:
- Efgartigimod PH20 SC: Patients randomized to receive weekly administrations of efgartigimod PH20 until CRmin (complete remission on minimal prednisone therapy) or end of treatment period or early roll-over to the open-label extension study ARGX-113-1905. All participants received concurrent oral prednisone (or equivalent) at a starting dosage of 0.5 mg/kg/day. The dose of prednisone was adjusted according to recommendations as per protocol
- Placebo PH20 SC: Patients randomized to receive weekly administrations of placebo PH20 SC until CRmin (complete remission on minimal prednisone therapy) or end of treatment period or early roll-over to the open-label extension study ARGX-113-1905. All participants received concurrent oral prednisone (or equivalent) at a starting dosage of 0.5 mg/kg/day. The dose of prednisone was adjusted according to recommendations as per protocol
Period: Overall Study
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Started | 147 | 75
Completed | 104 | 46
Not Completed | 43 | 29
Not completed — Adverse Event | 3 | 2
Not completed — Withdrawal by Subject | 3 | 7
Not completed — Lost to Follow-up | 2 | 0
Not completed — Physician Decision | 4 | 1
Not completed — Requires Prohibited Medication | 1 | 0
Not completed — lack of efficacy, geopolitical situation in Ukraine, flares after CRmin, SAE due to prednisone, etc | 30 | 19

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC | Total
Number analyzed (Participants) | 147 | 75 | 222
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.9 (12.55) | 52.3 (13.37) | 50.1 (12.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 73 | 42 | 115
  Male | 74 | 33 | 107
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 49 | 16 | 65
  Race: Black or African American | 1 | 2 | 3
  Race: White | 96 | 53 | 149
  Race: Other | 1 | 4 | 5
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 3 | 5 | 8
  Ethnicity: Not Hispanic or Latino | 144 | 70 | 214
Pemphigus Vulgaris (PV) [Count of Participants; unit: Participants] | 124 | 66 | 190
Pemphigus Foliaceus (PF) [Count of Participants; unit: Participants] | 23 | 9 | 32

OUTCOME MEASURES:

1. Primary Outcome: Number of Pemphigus Vulgaris (PV) Participants Who Achieve Complete Clinical Remission (CR) on Minimal Prednisone Therapy
Description: Proportion of participants with pemphigus vulgaris who had CRmin within 30 weeks, defined as the absence of new lesions and complete healing of established lesions while the participant was receiving prednisone at ≤10 mg/day for at least 8 weeks.
Time Frame: up to 30 weeks treatment period
Population: Randomized participants with pemphigus vulgaris (PV) who received at least part of a dose of efgartigimod PH20 SC or placebo PH20 SC. These participants also received prednisone with a starting dosage of 0.5 mg/kg/day. The dose of prednisone was adjusted per protocol
Measure: Count of Participants; unit: Participants
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 124 | 66
Participants | 44 | 20

2. Secondary Outcome: Number of Pemphigus Vulgaris (PV) and Pemphigus Foliaceus (PF) Participants Who Achieve Complete Clinical Remission (CR) on Minimal Prednisone Therapy Within 30 Weeks
Description: Proportion of participants with pemphigus vulgaris and pemphigus foliaceus who had CRmin within 30 weeks, defined as the absence of new lesions and complete healing of established lesions while the participant was receiving prednisone at ≤10 mg/day for at least 8 weeks.
Time Frame: up to 30 weeks treatment period
Population: Randomized participants with pemphigus vulgaris or pemphigus foliaceus who received at least part of a dose of efgartigimod PH20 SC or placebo PH20 SC. These participants also received prednisone with a starting dosage of 0.5 mg/kg/day. The dose of prednisone was adjusted per protocol.
Measure: Count of Participants; unit: Participants
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 147 | 75
Participants | 55 | 24

3. Secondary Outcome: Normalized Cumulative Prednisone Dose During the Treatment Period in Pemphigus Vulgaris Participants
Description: Normalized Cumulative prednisone dose (NCPD, mg/kg/day) is the average daily intake of all weight-adjusted prednisone doses received during the study, taking into account the number of days in study
Time Frame: Up to 30 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mg/kg/day
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 124 | 66
mg/kg/day | 0.416 (0.215) | 0.444 (0.232)

4. Secondary Outcome: Time to Complete Clinical Remission (CR) in Pemphigus Vulgaris Participants
Description: Time to complete remission (absence of new lesions and complete healing of established lesions) in participants with pemphigus vulgaris
Time Frame: Up to 30 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 124 | 66
days | 106 [79 to 161] | 120 [85 to 188]

5. Secondary Outcome: Time to Disease Control (DC) in Pemphigus Vulgaris (PV) Participants
Description: Time to disease control in participants with pemphigus vulgaris (Absence of new lesions and the start of healing of established lesions)
Time Frame: Up to 30 weeks
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 124 | 66
days | 16 [15 to 21] | 15 [8 to 17]

6. Secondary Outcome: Normalized Cumulative Prednisone Dose During the Treatment Period in Pemphigus Vulgaris and Pemphigus Foliaceus Participants
Description: as for outcome 3
Time Frame: Up to 30 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/kg/day
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 147 | 75
mg/kg/day | 0.403 (0.210) | 0.431 (0.225)

7. Secondary Outcome: Time to Complete Clinical Remission (CR) in Pemphigus Vulgaris and Pemphigus Foliaceus Participants
Description: Time to complete remission (absence of new lesions and complete healing of established lesions) in participants with pemphigus vulgaris and pemphigus foliaceus
Time Frame: Up to 30 weeks
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 147 | 75
days | 106 [84 to 142] | 113 [81 to 149]

8. Secondary Outcome: Time to Disease Control in Pemphigus Vulgaris and Pemphigus Foliaceus Participants
Description: Time to disease control in participants with pemphigus vulgaris and pemphigus foliaceus (Absence of new lesions and the start of healing of established lesions)
Time Frame: Up to 30 weeks
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
Number analyzed (Participants) | 147 | 75
days | 15 [15 to 17] | 15 [9 to 16]

ADVERSE EVENTS:
Time Frame: Up to 38 weeks
Description: Adverse events will be assessed at each participant visit. Treatment-emergent adverse events are reported in these tables. The adverse events were collected during the treatment period (up to 30 weeks) and in the follow-up period (up to 8 weeks) for participants who did not roll over to the OLE study (ARGX-113-1905).
Arm/Group | Efgartigimod PH20 SC | Placebo PH20 SC
All-Cause Mortality (participants affected / at risk) | 0/147 | 0/75
Serious Adverse Events (participants affected / at risk) | 18/147 | 10/75
Other Adverse Events (participants affected / at risk) | 113/147 | 47/75
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Efgartigimod PH20 SC (N=147) | Placebo PH20 SC (N=75)
ANAEMIA (Blood and lymphatic system disorders) | 0 | 1
TACHYCARDIA (Cardiac disorders) | 1 | 0
VISION BLURRED (Eye disorders) | 1 | 1
GASTRITIS EROSIVE (Gastrointestinal disorders) | 0 | 1
VOMITING (Gastrointestinal disorders) | 1 | 0
COVID-19 (Infections and infestations) | 2 | 2
COVID-19 PNEUMONIA (Infections and infestations) | 1 | 0
ERYSIPELAS (Infections and infestations) | 1 | 0
GASTROENTERITIS (Infections and infestations) | 1 | 0
PNEUMONIA (Infections and infestations) | 1 | 0
SKIN INFECTION (Infections and infestations) | 1 | 0
URINARY TRACT INFECTION (Infections and infestations) | 1 | 1
SPINAL COMPRESSION FRACTURE (Injury, poisoning and procedural complications) | 2 | 0
WEIGHT INCREASED (Investigations) | 1 | 0
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 | 1
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 0 | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPOPROTEINAEMIA (Metabolism and nutrition disorders) | 1 | 0
METABOLIC SYNDROME (Metabolism and nutrition disorders) | 0 | 1
SUPERFICIAL SPREADING MELANOMA STAGE UNSPECIFIED (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
HEADACHE (Nervous system disorders) | 0 | 1
GLOMERULONEPHRITIS (Renal and urinary disorders) | 1 | 0
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 1 | 0
DRUG ERUPTION (Skin and subcutaneous tissue disorders) | 1 | 0
PEMPHIGUS (Skin and subcutaneous tissue disorders) | 1 | 1
HYPERTENSION (Vascular disorders) | 2 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Efgartigimod PH20 SC (N=147) | Placebo PH20 SC (N=75)
INCREASED TENDENCY TO BRUISE (Blood and lymphatic system disorders) | 5 | 5
INJECTION SITE ERYTHEMA (General disorders) | 8 | 1
COVID-19 (Infections and infestations) | 17 | 3
NASOPHARYNGITIS (Infections and infestations) | 4 | 5
ORAL CANDIDIASIS (Infections and infestations) | 6 | 6
URINARY TRACT INFECTION (Infections and infestations) | 4 | 6
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 10 | 3
HYPERTRIGLYCERIDAEMIA (Metabolism and nutrition disorders) | 11 | 2
MYOPATHY (Musculoskeletal and connective tissue disorders) | 9 | 8
HEADACHE (Nervous system disorders) | 9 | 2
DEPRESSION (Psychiatric disorders) | 9 | 3
INSOMNIA (Psychiatric disorders) | 18 | 9
LEUKOCYTURIA (Renal and urinary disorders) | 4 | 4
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 7 | 6
HYPERTENSION (Vascular disorders) | 21 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-12-09): https://cdn.clinicaltrials.gov/large-docs/51/NCT04598451/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-22): https://cdn.clinicaltrials.gov/large-docs/51/NCT04598451/SAP_001.pdf